CLINICAL TRIAL: NCT05076058
Title: Effects of Tablets of Silybum Marianum, Pueraria Lobate and Salvia Miltiorrhiza on the Progression of Fatty Liver in Adults: a Double-blinded Randomized Placebo-controlled Clinical Trial
Brief Title: Effects of Tablets of Silybum Marianum, Pueraria Lobate and Salvia Miltiorrhiza on Fatty Liver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yu-ming Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K19-51000-043
Record Dates: First submitted 2021-09-10; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Fatty Liver Disease
Keywords: fatty liver; silybum marianum; Pueraria lobate; salvia miltiorrhiza
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — dan-shen root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo with the same appearance, taste, smell, and packing box to the experimental supplement was used. 118 serial numbers matched to each one participant, and corresponding to study arms (named as 1 or 2 on the tablet box), were used to replace the original label of supplement or placebo after randomization. The code of serial number corresponding to the group code (1 or 2) of tablets was kept by the PI, and will not be disclosed until the completion of all data collection. The group code corresponding to the two types of tablets was/will be kept by the producer till the completion of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Tablet name: tablet of silybum marianum, Pueraria lobate and salvia miltiorrhiza;
  Dosage: 1g/tablet, 3 tablets/time；
  Frequency: 2 times/day;
  Duration: 6 months
  Interventions: Dietary Supplement: Tablet of silybum marianum, Pueraria lobate and salvia miltiorrhiza
- Control group (Placebo Comparator): Tablet name: Placebo;
  Dosage: 1g/tablet, 3 tablets/time；
  Frequency: 2 times/day;
  Duration: 6 months
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Dietary Supplement: Tablet of silybum marianum, Pueraria lobate and salvia miltiorrhiza — Brand names: BY-HEALTH；
  Main contents (per 100g): silibinin 2g, salvianolic acid B 0.72g，Puerarin 0.68g
  Arms: Treatment group
Other: Placebo tablet — Brand names: BY-HEALTH；
  Main contents : starch
  Arms: Control group

SUMMARY:
Objectives: To examine the effects of tablets of silybum marianum, Pueraria lobate and salvia miltiorrhiza on the progression of fatty liver in patients with fatty liver.

Design: a double-blinded randomized placebo-controlled clinical trial.

Setting: community residents, Guangzhou city, South China.

Participants: a total 118 men and women (18-65 years), with BMI range of 24-30 kg/m2, and with fatty liver screened by ultrasound or MR at baseline.

Arms and Interventions: 118 participants were randomly allocated into two arms using a block randomization method. Experimental Arm: tablet of silybum marianum, Pueraria lobate and salvia miltiorrhiza, 3 tablets (1g each) twice a day for 6 months; Placebo Arm: placebo tablets, 3 tablets (1g each) twice a day for 6 months.

Outcome Measures: determined at baseline and at 6 months post treatment

1. Primary Outcome Measures: 1) proton density fat fraction of liver assessed by MR; 2) serum liver fibrosis biomarkers: type procollagen III N terminal peptide, hyaluronic acid, laminin, collagen type IV, and glycocholic acid; 3) NAFLD fibrosis score.
2. Secondary Outcome Measures: 1) serum liver function biomarkers: AST, ALT, GGT, ALP, total protein, and bile acids; 2) fasting blood lipids: total triglycerides, total cholesterol, HDL cholesterol and LDL cholesterol; 3) fasting serum glucose and insulin; 4) serum inflammatory factors (hsCRP and IL-6); 5) oxidative stress: SOD and MDA; and 6) body measurements and body fat mass.

Data Analyses: Mean changes in the above outcome measures from baseline to 6 months will be compared between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* BMI: 24-30 kg/m2
* Fatty liver, assessed by ultrasound or MR
* Had normal diet and normal daily life.

Exclusion Criteria:

* Hospital confirmed diseases of heart, liver (viral hepatitis, drug-induced liver injury, cirrhosis), kidney, brain, hematopoietic system，diabetes, immune system, and cancer；
* Taking medicine or supplements known to affect fatty liver, body fat;
* Body weight had changed more than 10% within the past 3 months;
* Physical or mental disabled to participate the trial;
* Compliance of tablet consumption is/was less than 80% in run-in period;
* Pregnant or lactating women, or intended pregnancy during the trial period;
* Be allergic to the proposed supplements；
* Attended or plan to attend other trial(s);
* Be unwell to sign the informed consent form, or have other conditions that be not suitable to attend the trial considered by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline proton density fat fraction of liver at 6 months | 0 and 6 months
  Proton density fat fraction of liver: measured using magnetic resonance (MR)
Change from baseline liver fibrosis biomarker (Type pro-collagen III N terminal peptide) at 6 months | 0 and 6 months
  Liver fibrosis biomarker 1: Type pro-collagen III N terminal peptide
Change from baseline liver fibrosis biomarker (hyaluronic acid) at 6 months | 0 and 6 months
  Liver fibrosis biomarker 2: hyaluronic acid
Change from baseline liver fibrosis biomarker (laminin) at 6 months | 0 and 6 months
  Liver fibrosis biomarker 3: laminin
Change from baseline liver fibrosis biomarker (collagen type IV) at 6 months | 0 and 6 months
  Liver fibrosis biomarker 4: Collagen type IV
Change from baseline liver fibrosis biomarker (glycocholic acid) at 6 months | 0 and 6 months
  Liver fibrosis biomarker 5: Glycocholic acid
Change from baseline NAFLD fibrosis score at 6 months | 0 and 6 months
  NAFLD fibrosis score: = -1.675 + 0.037 Age (yrs) + 0.094 BMI (kg/m2) + 1.13 impaired fasting glucose (IFG)/diabetes (yes = 1, no = 0) + 0.99 AST/ALT ratio - 0.013Platelet (*10E9/L) - 0.66 Albumin (g/dl)

SECONDARY OUTCOMES:
Change from baseline liver function biomarker (AST) at 6 months | 0 and 6 months
  Liver function biomarkers 1: AST
Change from baseline liver function biomarker (ALT) at 6 months | 0 and 6 months
  Liver function biomarkers 2: serum ALT
Change from baseline liver function biomarker (GGT) at 6 months | 0 and 6 months
  Liver function biomarkers 3: serum gamma-glutamyl transpeptidase (GGT)
Change from baseline liver function biomarker (total protein) at 6 months | 0 and 6 months
  Liver function biomarkers 4: serum total protein
Change from baseline liver function biomarker (ALP) at 6 months | 0 and 6 months
  Liver function biomarkers 5: serum alkaline phosphatase (ALP)
Change from baseline liver function biomarker (bile acids) at 6 months | 0 and 6 months
  Liver function biomarkers 6: serum bile acids
Change from baseline fasting blood lipid (TG) at 6 months | 0 and 6 months
  Fasting blood lipid 1: serum triglycerides
Change from baseline fasting blood lipid (TC) at 6 months | 0 and 6 months
  Fasting blood lipid 2: serum total cholesterol
Change from baseline fasting blood lipid (HDL-C) at 6 months | 0 and 6 months
  Fasting blood lipid 3: serum high-density lipoprotein cholesterol (HDL-C)
Change from baseline fasting blood lipid (LDL-C) at 6 months | 0 and 6 months
  Fasting blood lipid 4: serum low-density lipoprotein cholesterol (LDL-C)
Change from baseline fasting blood glucose at 6 months | 0 and 6 months
  Fasting blood glucose: serum glucose
Change from baseline fasting blood insulin at 6 months | 0 and 6 months
  Fasting blood insulin: serum insulin
Change from baseline systolic blood pressure at 6 months | 0 and 6 months
  Blood pressure: systolic blood pressure
Change from baseline diastolic blood pressure at 6 months | 0 and 6 months
  Blood pressure: diastolic blood pressure
Change from baseline Inflammatory factor (hsCRP ) at 6 months | 0 and 6 months
  Inflammatory factor 1: serum high sensitivity C reactive protein (hsCRP)
Change from baseline Inflammatory factor (IL-6) at 6 months | 0 and 6 months
  Inflammatory factor 2: serum IL-6
Change from baseline oxidative stress (SOD) at 6 months | 0 and 6 months
  Oxidative stress biomarker 1: serum SOD
Change from baseline oxidative stress (MDA) at 6 months | 0 and 6 months
  Oxidative stress biomarker 2: serum malondialdehyde (MDA)
Change from baseline fat mass at 6 months | 0 and 6 months
  Fat mass (FM): FM (kg) at total body and sub-regions determined by a dual energy x-ray absorptiometry (DXA)
Change from baseline percentage fat mass at 6 months | 0 and 6 months
  Percentage Fat mass (%FM): %FM (%) at total body and sub-regions determined by DXA

OTHER OUTCOMES:
Change from baseline body weight at 6 months | 0 and 6 months
  Body measurement 1: Body weight (in kg)
Change from baseline body height at 6 months | 0 and 6 months
  Body measurement 2: Body height (in cm)
Change from baseline waist circumference at 6 months | 0 and 6 months
  Body measurement 3: Waist circumference (in cm)
Change from baseline hip circumference at 6 months | 0 and 6 months
  Body measurement 4: hip circumference (in cm)
Change from baseline anxiety score at 6 months | 0 and 6 months
  Anxiety Score: assessed by a Self Rating Anxiety Scale (SAS).the minimum and maximum values: 25-100 points. Higher scores mean worse outcome.
Number of treated events related to supplements between baseline to 6 months | 0 and 6 months
  Adverse/side effects: Assessed by using questionnaire of medical history, medication use, symptoms.
Percentage of the interventional supplements consumed between baseline to 6 months | at 6 months
  Compliance assessment: Assessed by counting the number of remaining supplemental tablets at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li BY, Xi Y, Liu YP, Wang D, Wang C, Chen CG, Fang XH, Li ZX, Chen YM. Effects of Silybum marianum, Pueraria lobate, combined with Salvia miltiorrhiza tablets on non-alcoholic fatty liver disease in adults: A triple-blind, randomized, placebo-controlled clinical trial. Clin Nutr ESPEN. 2024 Oct;63:2-12. doi: 10.1016/j.clnesp.2024.06.003. Epub 2024 Jun 10. PMID 38879879